CLINICAL TRIAL: NCT05469178
Title: Phase 1b/2a Safety and Tolerability Study of Bemcentinib With Pembrolizumab/Carboplatin/Pemetrexed in Subjects With Untreated Advanced or Metastatic Non-squamous Non-small Cell Lung Cancer (NSCLC) Without/With a STK11 Mutation
Brief Title: A Clinical Study of Bemcentinib With Standard of Care Chemoimmunotherapy in Untreated Advanced/Metastatic Non-small Cell Lung Cancer Patients With a Mutation in the STK11 Gene
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: BerGenBio ASA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGBC016; 2024 511007 41 00 (EU CTIS Number); U1111-1312-8770 (Other: Universal Trial Number)
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — bemcentinib; pembrolizumab; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1b Cohort 1: Bemcentinib 75 mg (Experimental): Participants with previously untreated locally advanced (Stage IIIb/IIIc)/metastatic (Stage IV) non-squamous NSCLC without actionable mutations will receive bemcentinib 75 mg once daily until a reason for discontinuation has been met or for up to 2 years, whichever occurs first along with CIT (pembrolizumab infusion followed by pemetrexed and carboplatin).
  Interventions: Drug: Bemcentinib; Drug: Pembrolizumab; Drug: Pemetrexed; Drug: Carboplatin
- Phase 1b Cohort 2: Bemcentinib 100 mg (Experimental): Participants with previously untreated locally advanced (Stage IIIb/IIIc)/metastatic (Stage IV) non-squamous NSCLC without actionable mutations will receive bemcentinib 100 mg once daily until a reason for discontinuation has been met or for up to 2 years, whichever occurs first along with CIT (pembrolizumab infusion followed by pemetrexed and carboplatin).
  Interventions: Drug: Bemcentinib; Drug: Pembrolizumab; Drug: Pemetrexed; Drug: Carboplatin
- Phase 1b Cohort 3: Bemcentinib 150 mg (Experimental): Participants with previously untreated locally advanced (Stage IIIb/IIIc)/metastatic (Stage IV) non-squamous NSCLC without actionable mutations will receive bemcentinib 150 mg once daily until a reason for discontinuation has been met or for up to 2 years, whichever occurs first along with CIT (pembrolizumab infusion followed by pemetrexed and carboplatin).
  Interventions: Drug: Bemcentinib; Drug: Pembrolizumab; Drug: Pemetrexed; Drug: Carboplatin
- Phase 2a Expansion Cohort: Bemcentinib 100 mg (as the dose determined from Phase 1b) (Experimental): Participants with previously untreated advanced (Stage IIIb/IIIc)/metastatic (Stage IV) non-squamous NSCLC having a serine/threonine kinase 11 (STK11) mutation as identified by Next Generation Sequencing (NGS) and without actionable mutations will receive bemcentinib second dose, at RP2D identified in Phase 1b, once daily until a reason for discontinuation has been met or for up to 2 years, whichever occurs first along with CIT (pembrolizumab infusion followed by pemetrexed and carboplatin).
  Interventions: Drug: Bemcentinib; Drug: Pembrolizumab; Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: Bemcentinib — Bemcentinib capsules will be administered daily orally.
Drug: Pembrolizumab — Pembrolizumab will be administered as an intravenous (IV) infusion as part of CIT every 3 weeks.
Drug: Pemetrexed — Pemetrexed will be administered as an IV infusion as part of CIT every 3 weeks.
Drug: Carboplatin — Carboplatin will be administered as an IV infusion as part of CIT every 3 weeks up to 4 cycles. Each cycle = 21 days.

SUMMARY:
The primary purpose of this study is to determine the safety and tolerability of the combination of bemcentinib with chemo-immunotherapy (CIT) to identify the recommended phase 2 dose (RP2D) when administered as first line (1L) treatment in participants with locally advanced (Stage IIIb/IIIC) or metastatic (Stage IV) non-squamous NSCLC with no actionable mutations and to determine the anti-tumor activity of the combination of bemcentinib with CIT when administered as 1L treatment in participants with locally advanced (Stage IIIb/IIIc) or metastatic (Stage IV) non-squamous NSCLC with serine/threonine kinase 11 (STK11) mutation and no actionable mutations.

ELIGIBILITY:
Main Inclusion Criteria:

* Histologically-confirmed or cytologically confirmed diagnosis of advanced (Stage IIIb/IIIc) or metastatic (Stage IV) (AJCC Edition 8) non-squamous NSCLC not amenable to curative therapy, irrespective of PD-L1 status and without actionable mutations (Phase 1b) targetable with first-line treatment.
* Histologically-confirmed or cytologically confirmed diagnosis of stage of advanced (Stage IIIb/IIIC) or metastatic (Stage IV) (AJCC, Edition 8) non-squamous NSCLC with STK11 mutation, not amenable to curative therapy, irrespective of PD-L1 status and without actionable mutations (phase 2a) targetable with first-line treatment.
* Have not received prior systemic treatment for their advanced/metastatic NSCLC
* Have measurable disease per RECIST 1.1 as assessed by the investigator

Main Exclusion Criteria:

* Has received any prior chemotherapy or biological therapy for locally advanced (Stage IIIb/IIIc) or metastatic (Stage IV) adenocarcinoma of the lung
* Received radiation therapy within 2 weeks prior to starting study treatment or has not recovered (i.e. <=Grade 1 at baseline) from AEs due to a previous radiation therapy
* Major surgery within 28 days prior to start of study treatment and failure to have recovered adequately from the complications of the surgery/intervention prior to the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (7):
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - University of Chicago, Chicago, Illinois
  - Marlene and Stewart Greenebaum Comprehensive Cancer Center, University of Maryland, Baltimore, Maryland
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Duke University Medical Center - Duke Cancer Center, Durham, North Carolina
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
- France (4):
  - Hôpital prive du Confluent SAS, Departement d'oncologie, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hôpital Europeen Georges Pompidou (HEGP), Service de cancérologie, Paris
  - Institut Gustave Roussy, Service de médecine, Villejuif
- Greece (4):
  - Henry Dunant Hospital Center, 4th Oncology Department, Athens
  - Sotiria General Hospital of Chest Diseases, 3rd Department of Internal Medicine, Oncology Unit, Athens
  - General Hospital of Athens Alexandra, Department of the Clinical Therapeutics, Medical Oncology Unit, Athens
  - University General Hospital of Larissa, Oncology Clinic, Larissa
- Hungary (3):
  - Semmelweis University- Department of Pulmonology, Budapest
  - Orszagos Koranyi Pulmonologiai Intezet, Budapest
  - Fejer County St. Gyorgy Hospital, Székesfehérvár
- Italy (4):
  - Azienda Ospedaliero-Universitaria Policlinico S. Orsola-Malpighi, Bologna
  - Ospedale San Luca, Lucca
  - IRCCS - Istituto Europeo di Oncologia IEO, Milan
  - IFO Regina Elena, Rome
- Poland (4):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, II Klinika Chorob Pluc, raka płuca i chorób wewnętrznych, Bialystok
  - Instytut Centrum Zdrowia Matki Polki (ICZMP), Lodz
  - Uniwersytecki Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - MedPolonia Sp z oo, Poznan
- Spain (8):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - MD Anderson Cancer Center, Oncology service, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Fundacion Instituto Valenciano de Oncologia (FIVO), Valencia
  - Hospital Clinico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment was undertaken across 7 planned countries: USA, France, Greece, Hungary, Italy, Poland & Spain. Of these countries, 5 countries enrolled participants: USA (10 participants), France (5 participants), Greece (3 participants), Italy (2 participants) & Spain (6 participants). The recruitment process began in March 2023 and concluded in February 2025. 65 participants were screened in order to successfully recruit 26 participants.
Pre-assignment Details: Participants were screened to the inclusion/exclusion criteria of the protocol. The following assessments were performed: Informed Consent, Demographics, Medical/Surgical History including NSCLC diagnosis and prior anticancer treatments, Pregnancy/FSH, ECOG performance score, Vital signs, Physical examination, Echocardiogram, Laboratory Safety Testing, ECG, Tumour imaging/sampling and biopsies & blood sampling for genomic DNA/serum biomarkers.
Groups:
- Phase 2a Expansion Cohort: Bemcentinib 100 mg (as the dose determined from Phase 1b): Participants with previously untreated advanced (Stage IIIb/IIIc)/metastatic (Stage IV) non-squamous NSCLC having a serine/threonine kinase 11 (STK11) mutation as identified by Next Generation Sequencing (NGS) and without actionable mutations will receive bemcentinib, at RP2D identified in Phase 1b, once daily until a reason for discontinuation has been met or for up to 2 years, whichever occurs first along with CIT (pembrolizumab infusion followed by pemetrexed and carboplatin).
  Bemcentinib: Bemcentinib capsules will be administered daily orally.
  Pembrolizumab: Pembrolizumab will be administered as an intravenous (IV) infusion as part of CIT every 3 weeks.
  Pemetrexed: Pemetrexed will be administered as an IV infusion as part of CIT every 3 weeks.
  Carboplatin: Carboplatin will be administered as an IV infusion as part of CIT every 3 weeks up to 4 cycles. Each cycle = 21 days.
Period: Overall Study
Arm/Group | Phase 1b Cohort 1: Bemcentinib 75 mg | Phase 1b Cohort 2: Bemcentinib 100 mg | Phase 1b Cohort 3: Bemcentinib 150 mg | Phase 2a Expansion Cohort: Bemcentinib 100 mg (as the dose determined from Phase 1b)
Started | 3 | 3 | 4 | 16
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 4 | 16
Not completed — Death | 1 | 1 | 3 | 6
Not completed — Lack of Efficacy | 2 | 2 | 1 | 10

BASELINE CHARACTERISTICS:
Population: This analysis population includes all 26 enrolled participants.
Groups:
- Phase 1b Cohort 1: Bemcentinib 75 mg: Participants with previously untreated locally advanced (Stage IIIb/IIIc)/metastatic (Stage IV) non-squamous NSCLC without actionable mutations received oral bemcentinib 75 mg once daily until a reason for discontinuation had been met or for up to 2 years, whichever occurred first along with CIT (pembrolizumab infusion followed by pemetrexed and carboplatin). CIT was administered on day 1 of 21-day cycles via intravenous (IV) infusions and comprised pembrolizumab, pemetrexed, and carboplatin. Carboplatin was administered for a maximum of 4 cycles only.
- Phase 1b Cohort 2: Bemcentinib 100 mg: Participants with previously untreated locally advanced (Stage IIIb/IIIc)/metastatic (Stage IV) non-squamous NSCLC without actionable mutations received oral bemcentinib 100 mg once daily until a reason for discontinuation had been met or for up to 2 years, whichever occurred first along with CIT (pembrolizumab infusion followed by pemetrexed and carboplatin). CIT was administered on day 1 of 21-day cycles via intravenous (IV) infusions and comprised pembrolizumab, pemetrexed, and carboplatin. Carboplatin was administered for a maximum of 4 cycles only.
- Phase 1b Cohort 3: Bemcentinib 150 mg: Participants with previously untreated locally advanced (Stage IIIb/IIIc)/metastatic (Stage IV) non-squamous NSCLC without actionable mutations received oral bemcentinib 150 mg once daily until a reason for discontinuation had been met or for up to 2 years, whichever occurred first along with CIT (pembrolizumab infusion followed by pemetrexed and carboplatin). CIT was administered on day 1 of 21-day cycles via intravenous (IV) infusions and comprised pembrolizumab, pemetrexed, and carboplatin. Carboplatin was administered for a maximum of 4 cycles only.
- Phase 2a Expansion Cohort: Bemcentinib 100 mg (as the Dose Determined From Phase 1b): Participants with previously untreated advanced (Stage IIIb/IIIc)/metastatic (Stage IV) non-squamous NSCLC having a serine/threonine kinase 11 (STK11) mutation as identified by Next Generation Sequencing (NGS) and without actionable mutations will receive bemcentinib, at RP2D identified in Phase 1b, once daily until a reason for discontinuation has been met or for up to 2 years, whichever occurs first along with CIT (pembrolizumab infusion followed by pemetrexed and carboplatin). CIT was administered on day 1 of 21-day cycles via intravenous (IV) infusions and comprised pembrolizumab, pemetrexed, and carboplatin. Carboplatin was administered for a maximum of 4 cycles only.
- Total: Total of all reporting groups
Arm/Group | Phase 1b Cohort 1: Bemcentinib 75 mg | Phase 1b Cohort 2: Bemcentinib 100 mg | Phase 1b Cohort 3: Bemcentinib 150 mg | Phase 2a Expansion Cohort: Bemcentinib 100 mg (as the Dose Determined From Phase 1b) | Total
Number analyzed (Participants) | 3 | 3 | 4 | 16 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2 | 9 | 13
  >=65 years | 1 | 3 | 2 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.0 (26.66) | 71.0 (3.46) | 63.8 (7.14) | 61.2 (11.67) | 62.4 (15.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 0 | 3 | 5
  Male | 3 | 1 | 4 | 13 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 2 | 5
  Not Hispanic or Latino | 1 | 0 | 1 | 13 | 15
  Unknown or Not Reported | 1 | 1 | 3 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 2 | 1 | 4 | 14 | 21
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 0 | 1 | 4
Region of Enrollment [Number; unit: participants]
  Greece | 0 | 0 | 0 | 3 | 3
  United States | 2 | 2 | 1 | 5 | 10
  Italy | 0 | 0 | 0 | 2 | 2
  France | 1 | 1 | 3 | 0 | 5
  Spain | 0 | 0 | 0 | 6 | 6
Weight [Median (Full Range); unit: Kilograms] | 75.30 [63.0 to 81.6] | 82.00 [49.0 to 97.0] | 71.30 [61.2 to 82.2] | 70.50 [53.0 to 97.3] | 73.75 [49.0 to 97.0]
Height [Median (Full Range); unit: Centimetres] | 172.00 [170.0 to 188.0] | 165.00 [162.6 to 172.0] | 173.00 [168.0 to 184.0] | 171.00 [157.5 to 183.0] | 171.50 [162.6 to 188.0]

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose Limiting Toxicity (DLT)
Description: DLT graded using NCI CTCAE Version 5.0 based on the Investigator assessment.
Time Frame: Cycle 1 (the first 21 days of treatment)
Population: This analysis population included all 10 participants who were enrolled into Phase 1b of the study and completed at least one cycle of treatment for evaluation of DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Cohort 1: Bemcentinib 75 mg | Phase 1b Cohort 2: Bemcentinib 100 mg | Phase 1b Cohort 3: Bemcentinib 150 mg
Number analyzed (Participants) | 3 | 3 | 4
Participants | 0 | 0 | 0

2. Primary Outcome: Phase 2a: Objective Response Rate (ORR) at 6 Months
Description: ORR is defined as percentage of participants with complete response and partial response per RECIST 1.1.
Time Frame: 6 months
Population: This analysis population included all 16 participants who were enrolled into Phase 2a of the study and completed sufficient cycles of treatment up to the 6-month timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2a Expansion Cohort: Bemcentinib 100 mg (as the Dose Determined From Phase 1b)
Number analyzed (Participants) | 16
Participants | 0

3. Primary Outcome: Phase 2a: Objective Response Rate (ORR) at 12 Months
Description: ORR is defined as percentage of participants with complete response and partial response per RECIST 1.1.
Time Frame: 12 months
Population: This analysis population included all 16 participants who were enrolled into Phase 2a of the study and completed sufficient cycles of treatment up to the 12-month timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2a Expansion Cohort: Bemcentinib 100 mg (as the Dose Determined From Phase 1b)
Number analyzed (Participants) | 16
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from ICF signing until 30 days post the last treatment on study (approximately 1 year).
Description: All reported adverse events were mapped to standard MedDRA coding terms, grouped by system organ class and preferred term and tabulated by treatment cohorts.
Arm/Group | Phase 1b Cohort 1: Bemcentinib 75 mg | Phase 1b Cohort 2: Bemcentinib 100 mg | Phase 1b Cohort 3: Bemcentinib 150 mg | Phase 2a Expansion Cohort: Bemcentinib 100 mg (as the Dose Determined From Phase 1b)
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 3/4 | 6/16
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 1/4 | 6/16
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b Cohort 1: Bemcentinib 75 mg (N=3) | Phase 1b Cohort 2: Bemcentinib 100 mg (N=3) | Phase 1b Cohort 3: Bemcentinib 150 mg (N=4) | Phase 2a Expansion Cohort: Bemcentinib 100 mg (as the Dose Determined From Phase 1b) (N=16)
Claudication in Peripheral Vascular Disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Intermittent Claudication
Embolic Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (4) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Pyelonephritis E.coli Urinary Tract Infection
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (4) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelets Count Decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Weight Loss (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Weight Decreased
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Mucosal Inflammation
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Digestive Bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Upper Gastrointestinal Haemorrhage
Enterococcus Faecalis Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epigastralgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Abdominal Pain Upper
Secondary Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Secondary Adrenocortical Insufficiency
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White Blood Cells Decrease (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial Fibrillation With RVR (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bowel Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombolic Event - Right Ventricle (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Embolism
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b Cohort 1: Bemcentinib 75 mg (N=3) | Phase 1b Cohort 2: Bemcentinib 100 mg (N=3) | Phase 1b Cohort 3: Bemcentinib 150 mg (N=4) | Phase 2a Expansion Cohort: Bemcentinib 100 mg (as the Dose Determined From Phase 1b) (N=16)
Alanine Aminotransferase Increased (Investigations) | 1 (2) | 1 (2) | 3 (6) | 4 (6)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 5 (9)
Dry Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea on Exertion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythematous Lesions of the Anterior Face, Torso and Dorsal Root and Legs, Pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Erythema
Fatigue (General disorders) | 2 (3) | 1 (3) | 1 (1) | 1 (1)
Fever (General disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (4) — Pyrexia
Inappetence (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 2 (3) | 4 (8) — Decreased Appetite
Large Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (6) | 2 (6) | 4 (12) | 2 (4)
Neutropenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 1 (2) | 3 (5)
Acid Reflux (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) — Gastrooesophageal Reflux Disease
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Bilateral Leg Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Pain in Extremity
Claudication in Peripheral Vascular Disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Intermittent Claudication
Constipation (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1) | 4 (4)
Hand Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Pruritus
Head Pain (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Headache
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Short of Breath (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (4) | 2 (5) | 0 (0) — Dyspnoea
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swollen Legs (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Peripheral Swelling
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (7) | 4 (10) | 1 (2)
Embolic Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Embolic Stroke
Feeling Frail (General disorders) | 2 (2) | 0 (0) | 2 (2) | 4 (4) — Asthenia
Generalised Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Pollakiuria
Worsening Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Worsening of Prostatic Hyperplasia with Urinary Frequency (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Benign Prostatic Hyperplasia
Arthralgias (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 3 (4) | 3 (3)
Bronchial Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chronic Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Lower Limb Edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle Pain in Arms and Thighs (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Myalgia
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis E.coli Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Serious Otitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Ear Infection
Unknown Allergic Reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Hypersensitivity
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (5) | 5 (6)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Creatinine Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (4) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Average QTCF Greater than 450ms (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Electrocardiogram Qt Prolonged
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis Immunomediated (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema Face and Chest (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase Increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Melanoderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis Oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) — Stomatitis
Seborrheic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trunk Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Watery Eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Lacrimation
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deterioration of General Condition (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hand Foot Syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Palmar-Plantar Erythrodysaesthesia Syndrome
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelets Count Decreased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 3 (6)
Skin Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight Loss (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Bulbar Gastric Ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophil Count Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Increased Alkaline Phosphatase (Investigations) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Increased Basophils (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased Lactate Dehydrogenase (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased Neutrophils (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Monocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-Pruritic Maculopapular Skin Lesions of the Extremities (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet Count Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety Worsening (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT Corrected Interval Prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (5) | 2 (2)
Neutrophil Count Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White Blood Cells Decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 3 (4)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amylase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dry Eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper and Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Body Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema in Left Lower Extremity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Oedema Peripheral
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left Femoral Oncologic Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral Pain due to Mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Stomatitis
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal Insufficiency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal Ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Feet and Hand Edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Oedema Peripheral
Gamma Glutamyltransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Influenza A Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Foot Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Digestive Bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Upper Gastrointestinal Haemorrhage
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (10)
Bilateral and Dorsal Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosity (Site Unknown) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Mucosal Inflammation
Skin Rash on the Chest (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Entercoccus Faecalis Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epigastralgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Abdominal Pain Upper
Secondary Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lymphocytes Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Malleolus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Thyroid Nodule (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cranial Theca Pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Headache
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Left Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — Arthralgia
Right Arm Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Rash (Lateral Thigh) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blurred Vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial Fibrillation with RVR (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Grade 3 Lymphocyte Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Hypoxic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bowel Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
International Normalised Ratio Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impaired Skin Integrity around Nail Bed (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombolic Event - Right Ventricle (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Embolism

LIMITATIONS AND CAVEATS:
The study was terminated early due to lack of efficacy, therefore the study enrolled a smaller than planned number of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure agreement outlines that PIs are not to disclose study results without prior discussion with the study Sponsor

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT05469178/Prot_SAP_000.pdf